CLINICAL TRIAL: NCT05937750
Title: A Prospective, Post-authorisation Long-term Follow-up Trial of Patients Previously Treated With Imlifidase Prior to Kidney Transplantation, Including a Non-comparative Concurrent Reference Cohort
Brief Title: A Long-term Follow-up Trial of Patients Previously Treated With Imlifidase Prior to Kidney Transplantation and a Non-comparative Transplanted Patient Group
Acronym: PAES-LTFU
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-HMedIdeS-20
Record Dates: First submitted 2023-06-13; First posted 2023-07-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Long Term Efficacy and Safety
Keywords: Renal transplantation; Kidney transplantation
MeSH Terms: interventions — phenyl-2-aminoethyl sulfide

STUDY DESIGN:
Intervention Model Description: This is a long-term follow-up trial following an open-label, non-randomized trial in highly sensitized adult kidney transplant patients with positive crossmatch (XM) against an available deceased donor.
  The rational for the main trial, 20-HMedIdeS-19 (PAES), being non-randomized is that no other effective or approved desensitization protocol exists in deceased-donor kidney transplantation that would provide a suitable control. A non-comparative concurrent reference cohort from participating sites was included to address differences in-site practice and experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imlifidase (Experimental): Imlifidase administered in the 20-HMedIdeS-19 (PAES) study
  Interventions: Drug: Imlifidase administered in the 20-HMedIdeS-19 (PAES) study
- Non-Comparative Concurrent Reference Cohort (Experimental): Best available treatment administered in the 20-HMedIdeS-19 (PAES) study
  Interventions: Other: Best available treatment administered in the 20-HMedIdeS-19 (PAES) study

INTERVENTIONS:
Drug: Imlifidase administered in the 20-HMedIdeS-19 (PAES) study — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly selective towards IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc-fragment and efficiently neutralizes Fc-mediated activities of IgG.
  Other Names: IdeS; HMED-IdeS; Idefirix
  Arms: Imlifidase
Other: Best available treatment administered in the 20-HMedIdeS-19 (PAES) study — Normal transplantation routine Transplantation and pre- and post-transplantation therapies in accordance with the clinic's normal transplantation routine.
  Arms: Non-Comparative Concurrent Reference Cohort

SUMMARY:
A prospective, post-authorisation long-term follow-up trial of patients previously treated with imlifidase prior to kidney transplantation, including a non-comparative concurrent reference cohort.

DETAILED DESCRIPTION:
This is a long-term follow-up trial to the post-authorisation efficacy and safety (PAES) trial (trial 20-HMedIdeS-19). The trial will include patients who participated in the PAES trial and were transplanted with a new kidney after treatment with imlifidase (trial drug) or standard of care medication. Imlifidase is a medicine used to prevent the body from rejecting a newly transplanted kidney and is used before transplantation in adults who have antibodies against the donor kidney and are considered 'highly sensitised' based on a positive crossmatch test.

The purpose of this follow-up trial is to fulfil requirements from the European Medicines Agency (EMA) to continue to evaluate efficacy (kidney function) and safety (side effects) over time, for the patients who were transplanted with a new kidney in the PAES trial. The patients will be followed for up to 5 years after transplantation in the PAES trial to collect valuable long-term data.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent obtained before any trial-related procedures
* Willingness and ability to comply with the protocol
* Previously transplanted in the clinical trial 20-HmedIdeS-19 (PAES)

Exclusion Criteria:

* Inability by the judgment of the investigator to participate in the trial for other reasons

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Graft failure-free survival (%) up to 5 years after imlifidase enabled transplantation (imlifidase cohort only) | 5-years after transplantation
  Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients not undergoing transplantation will be censored at time zero (i.e. at entry into the PAES trial). Transplanted patients not having an event (graft failure or death) will be censored at the last known date being alive and having a functioning graft.
  The 5-year graft failure-free survival rates will be estimated using the Kaplan-Meier estimator. Time from enrolment to the first of death or graft failure will be used as time variable.

SECONDARY OUTCOMES:
Graft failure-free survival (%) up to 5 years after transplantation (non-comparative concurrent reference cohort only) | 5-years after transplantation
  Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients not undergoing transplantation will be censored at time zero (i.e. at entry into the PAES trial). Transplanted patients not having an event (graft failure or death) will be censored at the last known date being alive and having a functioning graft.
  The 5-year graft failure-free survival rates will be estimated using the Kaplan-Meier estimator. Time from enrolment to the first of death or graft failure will be used as time variable.
Graft failure-free survival (%) up to 2 and 3 years after transplantation | 2 and 3-years after transplantation
  Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients not undergoing transplantation will be censored at time zero (i.e. at entry into the PAES trial). Transplanted patients not having an event (graft failure or death) will be censored at the last known date being alive and having a functioning graft.
  The 2 and 3-year graft failure-free survival rates will be estimated using the Kaplan-Meier estimator. Time from enrolment to the first of death or graft failure will be used as time variable.
Renal function as evaluated by estimated Glomerular Filtration Rate (eGFR) and serum/plasma creatinine levels | 2, 3, and 5-years after transplantation
  Kidney function assessed by eGFR and serum/plasma creatinine will be summarised over 5 years for the imlifidase group and the reference cohort.
  eGFR is a measure of kidney function. The serum/plasma creatinine levels will be analysed and eGFR will be calculated according to the modification of diet in renal disease (MDRD) equation.
  Reduced kidney function is characterised by a decreased eGFR value. For patients in the imlifidase group who are not successfully transplanted, or for any enrolled patients without a functioning graft, their eGFR values will be set to 0 mL/min.
Patient survival (%) after transplantation | 2, 3, and 5-years after transplantation
  Patient survival up to 2, 3 and 5 years, respectively, will be assessed for the imlifidase group and the reference cohort.
  The 2, 3, and 5-year patient survival rates will be extracted from Kaplan-Meier curves.
Graft survival (%) after transplantation | 2, 3, and 5-years after transplantation
  Graft survival up to 2, 3 and 5 years, respectively, will be assessed for the imlifidase group and the reference cohort.
  Graft survival will be presented with Kaplan-Meier curves. Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients who die will be censored at time of death.
Human Leukocyte Antigen (HLA)/Donor Specific Antibodies (DSA) levels (imlifidase cohort only) | 2, 3, and 5-years after transplantation
  HLA antibodies will be analysed using an IgG single antigen solid-phase immunoassay for class I and class II (SAB-HLA).
  Donor specific antibodies (DSAs) are identified by using the human leukocyte antigen (HLA) profile data from the donor and the recipient to identify HLA-mismatches.
  The mean fluorescence intensity (MFI) will be summarized for all DSAs with an MFI of ≥1000 at any time during the trial (or the PAES trial).
Anti-drug antibody (ADA) levels (imlifidase cohort only) | 2, 3, and 5-years after transplantation
  Determination of anti-imlifidase IgG (ADA) concentration in serum will be performed centrally using a customised ImmunoCAP to evaluate imlifidase long-term immunogenicity.
Proportion of patients (%) with biopsy- and serology (DSA)-confirmed Antibody Mediated Rejections (AMRs) | 2, 3, and 5-years after transplantation
  For-cause biopsies will be obtained to confirm diagnosis for suspected AMRs in both treatment arms.
  The biopsies will be analysed locally and centrally and evaluated according to Banff criteria version 2017 or later.
Proportion of patients (%) with biopsy confirmed Cell-Mediated Rejections (CMRs) | 2, 3, and 5-years after transplantation
  For-cause biopsies will be obtained to confirm diagnosis for suspected CMRs in both treatment arms.
  The biopsies will be analysed locally and centrally and evaluated according to Banff criteria version 2017 or later.
Treatment of graft rejections | 2, 3, and 5-years after transplantation
  The number of graft rejection episodes treated with dialysis will be recorded
Treatment of graft rejection | 2, 3, and 5-years after transplantation
  The number of graft rejection episodes treated with plasmapheresis will be recorded
Treatment of graft rejection | 2, 3, and 5-years after transplantation
  The number of graft rejection episodes treated with medication will be recorded
Adverse events (AEs)/serious adverse events (SAEs) suspected to be related to imlifidase treatment (imlifidase cohort only) | 2, 3, and 5-years after transplantation
  AEs/SAEs suspected to be related to imlifidase treatment in the PAES trial will be recorded from the time of signed informed consent for participation in the trial until the last trial visit.
Use of immunosuppressive medication | 2, 3, and 5-years after transplantation
  The patient's use of immunosuppressive medications will be recorded for both cohorts from the time of signed informed consent for participation in the trial until the last trial visit.
Comorbidities | 2, 3, and 5-years after transplantation
  Information about comorbidities that are medically relevant and registered in the patient' medical record will be collected. Medically relevant comorbidities are infections, malignancy, diabetes mellitus and cardiovascular events.
Change in patient reported life participation | 2, 3, and 5-years after transplantation
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Social Health domain "Ability to participate in social roles & activities, PROMIS-SF-8a" will be used as a measure of the patients' health related quality of life.
  The questionnaire includes 8 questions about a persons ability to participate in different social activities and there are 5 different answers to choose from for each question: Never/Rarely/Sometimes/Usually/Always

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (13):
- Medizinische Universitaet Wien, Vienna, Austria
- Nephrology Clinic Vídeňská 1958/9, Prague, Czechia
- France (2):
  - Centre Hospitalier Universitaire (CHU) de Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume, Normandy
  - Hôpital Necker - Enfants Malades, Paris
- Azienda Ospedaliera di Padova, Padua, Italy
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus University Medical Center, Rotterdam
- Spain (4):
  - Hospital Del Mar, Servicio de Nefrología, Barcelona
  - Hospital Universitario del Vall d´Hebron, Barcelona
  - Unidad de Trasplante Renal, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- Sweden (2):
  - Karolinska University Hospital,, Huddinge, Stockholm County
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No